CLINICAL TRIAL: NCT01560013
Title: Brain Imaging Study on the Effects of Treatment With Naltrexone on Cue-induced Craving and Brain's Metabolic Changes in Alcohol and Cannabis-dependent Patients
Brief Title: The Effects of Treatment With Naltrexone in Alcohol and Cannabis-dependent Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112-10-TLV
Record Dates: First submitted 2010-06-03; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Alcohol-dependence
Keywords: Alcohol; naltrexone; cue reactivity; PET
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naltrexone (Experimental): Treatment with naltrexone for two months together with psycho-social support
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltrexone, oral 50 mg per day.
  Other Names: Revia

SUMMARY:
Alcohol dependence is a major health problem worldwide and recently in Israel and it has major health care costs. Cannabis dependence is also a major health issue and many cannabis users find it difficult to quit. Similar to dependence on heavy drugs, alcohol and cannabis-dependent patients find it difficult to quit drinking and smoking cannabis and they relapse to drinking alcohol and using cannabis during treatment. Craving for alcohol and cannabis and withdrawal during detoxification are major factors for relapse to drinking and using cannabis. The cue-exposure and priming paradigms have been used in order to induce craving for alcohol and cannabis in the laboratory. Several studies have delineated the brain mechanisms responsible for cue-induced craving for alcohol using functional Magnetic Resonance Imaging (fMRI), a method that can be useful in monitoring progress of treatment. A proven useful medication for treatment of alcohol dependence is the opiate antagonist naltrexone commonly used for treatment of opiate dependence. We have found that cannabis-dependent patients in treatment for cannabis dependence who also were heavy users of alcohol have dropped early from treatment.

DETAILED DESCRIPTION:
We propose to use naltexone to reduce craving for alcohol and cannabis in alcohol and cannabis-dependent patients. We also propose to use established techniques of priming and cue-exposure for alcoholic drinks and cannabis together with measures of [18F] Fluorodeoxyglucose (FDG) in Positron Emission Tomography (PET) imaging in 24 alcohol and cannabis-dependent patients before and after 35 day treatment with naltrexone. We predict that in those who will be successful in quitting alcohol drinking and using cannabis there would be a reduction in alcohol and cannabis cue-induced brain activity in the meso-limbic reward circuit that is responsible for craving for alcohol and cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependent patients both males and females age 22-64

Exclusion Criteria:

* subjects who are diagnosed as suffering from psychotic illness according to DSM-IV (Axis 1) (American Psychiatric Association, 1994) or with a history of CNS disease, a history of infection that might affect CNS (HIV, syphilis, cytomegalovirus, herpes), a history of head injury with loss of consciousness, history of other substance abuse taking psychoactive medications (shown by urine test). Abnormal liver test results (150% above average) will be excluded. Pregnancy is also an exclusion criterion, as radiation exposure is risky for the fetus.

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Verified abstinence from alcohol | 2 months
  Patients will be tested for alcohol at the end of treatment after 2 months

SECONDARY OUTCOMES:
Changes in subjective responses to alcohol-cue reactivity and brain's metabolic rates | At baseline and after treatment
  Alcohol and cannabis-dependent patients undergoing treatment with naltrexone will be assessed before and after treatment by the alcohol-cue exposure together with measures of the brain's metabolism using [18F] Fluoro-dioxyglucose (FDG) as the radiotracer in Positron Emission Tomography (PET) and subjective craving responses to the cues.

CONTACTS AND LOCATIONS:
Overall Officials: Aviv M Weinstein, Principal Investigator — TASMC Israel
Locations (1):
- Dept. of Nuclear Medicine, TASMC, Tel Aviv, Israel